CLINICAL TRIAL: NCT06801301
Title: Whole Body Vibration Versus Resisted Training on Strength of Quadriceps Post Lower Limb Burn.
Brief Title: Comparing Effects of Whole Body Vibration and Resisted Training on Quadriceps Strength After Lower Limb Burns
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Salah mohamed shafiek abuelfadl, Physiotherapy Specialist, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P.T.REC/012/002762
Record Dates: First submitted 2025-01-20; First posted 2025-01-30 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Lower Limb Burn; Muscle Weakness Condition
Keywords: Burn; Whole Body Vibration; Resisted Exercise; Isokinetic
MeSH Terms: conditions — Burns | interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- group A (Experimental): whole body vibration group
  Interventions: Device: whole body vibration
- group B (Active Comparator): resistance exercises
  Interventions: Other: Resistance Exercise

INTERVENTIONS:
Device: whole body vibration — Standing in different static positions or exercising on a vibrating platform.The mechanical stimuli of vibration transmitted to the body and stimulate muscle spindles which activate the alpha motor neurons and initiates muscle contractions comparable to the ''tonic vibration reflex. The effect of WBV on the neuromuscular properties of skeletal muscles and spinal mechanisms is demonstrated by a decreased electromechanical delay.
  Arms: group A
Other: Resistance Exercise — Resistance training as a mode of exercise to promote several health benefits, including improvements in the muscle mass and strength of healthy adults.Resistance training, where muscles are required to contract against an opposing load, has been shown to be a beneficial form of rehabilitation in clinical populations prone to muscle wasting, providing stimuli to increase protein synthesis and muscle mass.
  Arms: group B

SUMMARY:
Evaluate the therapeutic effect of Whole body vibration and Resistance training on strength of quadriceps post lower limb burn

DETAILED DESCRIPTION:
Study Design:

This randomized controlled trial will include 60 patients suffering from partial thickness burns. The patients will be randomly divided into two equal groups, with each group consisting of 30 patients.

Study Explanation:

A verbal explanation about the importance of the study, its procedures, main aims, and conceptual approach will be provided to every patient.

Study Procedures:

The procedures of this study will be divided into two main categories: evaluation procedures and treatment procedures.

Evaluation Procedures:

Evaluation will be conducted using isokinetic dynamometry for all patients both before and after the study.

Treatment Procedures:

First Group: Patients in the first group will receive whole body vibration therapy.

Second Group: Patients in the second group will undergo resisted exercises.

ELIGIBILITY:
Inclusion Criteria:

The subject selection will be according to the following criteria:

* Age range between 25-40 years.
* Male and female patients will participate in the study.
* All patients have burn of 30% to 40%.
* All patients have burn at lower limb
* All patients have second degree burn
* All patients have no chronic diseases.
* All patients enrolled to the study will have their informed consent

Exclusion Criteria:

The potential participants will be excluded if they meet one of the following criteria:

* Prosthesis;
* Any neurological, musculoskeletal,or other chronic disease
* Participation in an outside resistance training programs
* Recent fracture or bone injury
* Any medication that could affect strength adaptations and adversely affect the results of the study
* Previous brain injury
* Any disease affecting balance, vestibular or visual disorders
* History of epilepsy.
* Cardiac diseases.
* Burn of sole of foot.
* Exposed foot tendons.
* Severe osteopathy.
* Marked anemia (Ht<25%).
* Serious peripheral vessel disease
* Acute medical problem at study onset.

Ages: 25 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Increase in quadriceps muscle strength, assessed by an isokinetic dynamometer, which measures the peak torque of the quadriceps. | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Eman Mohamed Othman, doctoral degree, Study Director — Cairo University; Khadra Mohamed Ali, Doctoral degree, Study Chair — Cairo University; Ashraf El Sebaie Mohamed, doctoral, Study Director — Cairo University
Locations (1):
- Faculty of physical therapy cairo university, Cairo, Egypt, Egypt

IPD SHARING:
Plan to Share IPD: Yes